CLINICAL TRIAL: NCT07149246
Title: The Effect of a 6-month DiEtitian-TAILored Nutrition Intervention Compared to Usual Care in Patients With Critical Illness. A Single Center Prospective Intervention Study
Brief Title: The Effect of a 6-month Dietitian-tailored Nutrition Intervention to Patients With Critical Illness (DETAIL)
Acronym: DETAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Northern Norway Health Authority (Unknown); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Benjamin Kildal, Senior Consultant in Anesthesiology and Intensive Care, University Hospital of North Norway
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/882796 (REK); HNF1745-25 (Other Grant/Funding Number: Northern Norway Regional Health Authority)
Record Dates: First submitted 2025-08-05; First posted 2025-08-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: ICU Patients; Nutrition Intake; Critical Illness
Keywords: Nutrition; Energy intake; Protein intake; ICU; Dietitian
MeSH Terms: conditions — Critical Illness | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention)
- Nutrition intervention (Experimental): A 6-month Dietitian-tailored nutrition intervention
  Interventions: Other: Nutrition intervention

INTERVENTIONS:
Other: Nutrition intervention — Frequent follow-up from a dietitian during ICU and hospital stay, and after discharge, up to 6 months after ICU admission.
  Arms: Nutrition intervention

SUMMARY:
This research project aims to study the effect of optimal and individualised nutrition to patients with critical illness during the intensive care unit (ICU) and hospital admission, and until six months after admission. The investigators want to describe and compare the usual care with a dietitian-tailored nutrition care. The hypothesis is that dietitian-tailored nutrition care will result in a higher mean energy intake compared to usual care.

DETAILED DESCRIPTION:
The study will recruit patients with critical illness in one of two groups. Group one will receive standard nutrition care following the current local guidelines. Group two will receive frequent follow-up by a clinical dietitian from inclusion and until six months from admission. The dietitian will be responsible for the nutrition administered to the patient during hospital admission and will have consultations with the patients after discharge. The patients in group two will receive individualized nutrition care and recommendations.

In addition to outcome measures regarding nutrition, the patients can choose if they want to perform physical tests and blood tests as well, but that part of the study is optional. In both groups, outcome measures will be collected at day ten, 30, 90 and 180 days after admission to the ICU. The collection of data will occur even though the patients have been discharged from the hospital, either to their home or another health care facility.

The aim is to study the effect of optimal and individualised nutrition to patients with critical illness during the ICU and hospital admission, and until six months after admission. Firstly, the investigators want to describe the usual care and progression of the patients during the first six months after hospital admission. Secondly, the investigators want to see if frequent follow-up by a clinical dietitian can increase nutritional intake during the same period.

The hypothesis is that dietitian-tailored nutrition care will result in a higher mean energy intake compared to usual care, and that this will further impact other aspects, such as quality of life and physical function.

ELIGIBILITY:
Inclusion Criteria: Patients in intensive care who gives an informed consent and meet all of the following will be eligible:

1. Admitted to the intensive care unit for >48 hours.
2. At least 18 years of age
3. Have one or more organ system failure (respiratory,cardiovascular or renal) related to their acute illness defined as:

   a. PaO2/FiO2≤300 mm Hg) b. Currently on one or more continuous inotrope/vasopressor infusion which were started at least 4 hours ago at a minimum dose of: i. Norepinephrine≥0.1 mcg/kg/min ii. Epinephrine≥0.1 mcg/kg/min iii. Any dose of vasopressin iv. Milrinone>0.1 mcg/kg/min) c. Renal dysfunction defined as: i. Serum creatinine 2.0-2.9 times baseline or ii. Urine output 0.5 mL/kg/hour for ≥12 hours or iii. Currently receiving renal replacement therapy) d. Currently has an intracranial pressure monitor or ventricular drain in situ
4. Permanent living address in Norway

Exclusion Criteria: Patients will be excluded if:

1. Death is imminent in the next 96 hours or there is a current treatment limitation in place or the patient is unlikely to survive to 180 days due to underlying/chronic illness
2. Dialysis dependent chronic renal failure
3. Suspected or known pregnancy
4. Wheelchair user
5. Cognitive impairment in which intervention is considered not appropriate
6. Eating disorders -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean energy intake | Up to 6 months
  Mean energy intake from day 10 to the end of follow-up of 6 months.

SECONDARY OUTCOMES:
Protein intake | Up to 6 months
  Mean protein intake from day 10 to the end of follow-up of 6 months.
Nutrition intake | Day 10, day 30, day 90 and day 180
  Energy and protein intake on each measurement point, Energy and protein intake by location (intensive care unit and ward), Energy and protein intake delivered by nutrition therapy
Nutrition risk during overall follow-up | Baseline, day 10, day 30, day 90 and day 180
  Assessed with Nutrition Risk Screening 2002 (NRS-2002) at all measure time points, where the score 0-2 indicate no nutrition risk, and a score > 3 indicate nutrition risk.
Nutrition risk during ICU admission | ICU admission up to 6 months
  Assessed with the modified Nutrition Risk in Critically Ill (mNUTRIC) score, ranging from a minimum value of 0 and a maximum value of 9. 0-4 points indicate a low malnutrition risk, 5-9 points indicate patients at high nutrition risk which are the most likely to benefit from aggressive nutrition therapy.
Health related quality of life | Day 10, day 30, day 90 and day 180
  Assessed using the European Quality Of Life 5 Dimensions (EQ-5D) descriptive system. Each dimension has 5 levels ranging from no problems (1) to extreme problems (5), there is no overall score.
Self-rated health state | Day 10, day 30, day 90 and day 180
  Self-rated by the participants using the European Quality Of Life Visual Analogue Scale (EQ-VAS). The VAS ranges from "The worst health you can imagine" (0) to "The best health you can imagine" (100).
Frailty | Baseline, day 10, day 30, day 90 and day 180
  Assessed with clinical frailty scale (CFS), which is an ordinal scale with nine steps from very fit (1) to terminally ill (9).
Mobility | ICU admission up to 6 months
  Assessed during intensive care unit (ICU) admission using the 11-category ICU Mobility Scale, with 10 as the maximum value, where 0 indicate no activity and 10 indicate independent walking.
Weight | Baseline, day 10, day 30, day 90 and day 180
  Weight, Changes in weight between measurement points
Physical performance | Day 10, day 30, day 90 and day 180
  Changes in physical performance will be assessed using the Short Physical Performance Battery (SPPB). It consists of three tests; gait speed, balance test and a sit-to-stand test. The scores of the three tests are summarized, and the total score is ranging from 0 points to a maximum of 12 points. The score is divided in three levels of performance: low (0-6 points), medium (7-9 points), and high (10-12 points)
Hand grip strength | Day 10, day 30, day 90 and day 180
  Changes in hand grip strength assessed with a hand dynamometer
Body composition | Day 10, day 30, day 90 and day 180
  Changes in fat-free mass and lean mass assessed with bioelectrical impedance analysis (BIA).
Muscle mass | Baseline, day 10, day 30, day 90 and day 180
  Changes in muscle mass assessed with ultrasound
Resting energy expenditure | Day 10, day 30, day 90 and day 180
  Changes in resting energy expenditure measured with indirect calorimetry

OTHER OUTCOMES:
ICU stay | Up to 6 months
  Duration of intensive care unit (ICU) stay in survivors and non-survivors
Hospital stay | Up to 6 months
  Duration of hospital stay in survivors and non-survivors
Mortality | Up to 6 months
  Intensive care unit (ICU), in hospital and 30-day, 90-day and 6 months mortality
Effect of energy intake above 20 kcal/kg/dag | Day 10, day 30, day 90 and day 180
  Independent of group allocation, an analysis regarding all secondary outcome measures will be performed comparing participants with an energy intake of >20 kcal/kg/day with participants with <20 kcal/kg/day
Effect of energy intake above 25 kcal/kg/day | Day 10, day 30, day 90 and day 180
  Independent of group allocation, two analysis regarding all secondary outcome measures will be performed comparing participants with an energy intake of >25 kcal/kg/day with participants with <25 kcal/kg/day.
Cost per quality-adjusted life year | 6 months
  Cost per quality-adjusted life year (QALY)
Cost per life-year gained | 6 months
  Cost per life-year gained (LYG)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Benjamin Kildal, MD, PHD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient confidentiality. Parts of the data set may be available on reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT07149246/Prot_SAP_000.pdf